CLINICAL TRIAL: NCT01265173
Title: Comparison of Efficacy of Cefotaxime, Ceftriaxone, and Ciprofloxacin for the Treatment of Spontaneous Bacterial Peritonitis in Patients With Liver Cirrhosis
Brief Title: Comparison of Efficacy of Cefotaxime, Ceftriaxone, and Ciprofloxacin for the Treatment of SBP in Patients With LC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCCCSBP
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: SBP; Liver Cirrhosis
Keywords: SBP; liver cirrhosis; antibiotics
MeSH Terms: conditions — Liver Cirrhosis | interventions — Cefotaxime; Ceftriaxone; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cefotaxime (Active Comparator): iv 2G q 8hrs for general, dose titration if needed (eg.CKD)
  Interventions: Drug: Cefotaxime
- Ceftriaxone (Experimental): iv 2G q 24hrs
  Interventions: Drug: Ceftriaxone
- Ciprofloxacine (Experimental): iv 400mg q 12hrs for general, dose titration if needed (eg.CKD)
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Cefotaxime — 3 g
  Arms: Cefotaxime
Drug: Ceftriaxone — 2 g
  Arms: Ceftriaxone
Drug: Ciprofloxacin — 400 mg
  Arms: Ciprofloxacine

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is one of the most serious complications of liver cirrhosis. Mainstay of treatment for SBP is use of proper antibiotics. Although, several antibiotics including cefotaxime, ceftriaxone, or ciprofloxacin are being used, it is unclear which drug is most effective. Our aim of study is to compare the efficacy of the three current antibiotics for the treatment of SBP in patients with liver cirrhosis.

The primary hypothesis is that the efficacy of all the antibiotics will not significantly different. This is non-inferiority trial.

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is one of the most serious complications of liver cirrhosis. Mainstay of treatment for SBP is use of proper antibiotics. Although, several antibiotics including cefotaxime, ceftriaxone, or ciprofloxacin are being used, it is unclear which drug is most effective. Our aim of study is to compare the efficacy of the three current antibiotics for the treatment of SBP in patients with liver cirrhosis.

The primary hypothesis is that the efficacy of all the antibiotics will not significantly different. The expected success rates (infection resolution rates) are 83%, 87%, and 78% for cefotaxime, ceftriaxone, and ciprofloxacin. This is non-inferiority trial. The level of significance is 5%. The power of this stuy is 80%. Non-inferiority margin is 15%. Therefore 87 patients for each group are needed.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis patients with ascites
2. Ascitic fluid PMN cell count >250/mm3
3. Age: 16~70 years old

Exclusion Criteria:

1. Allergic to 3rd generation cephalosporin or quinolone
2. Antibiotics within 2 weeks
3. Open abdominal surgery within 4 weeks
4. Evidence of 2ndary peritonitis, intrabdominal hemorrhage, pancreatitis, Tb peritonitis, or peritoneal carcinomatosis
5. HCC with portal vein thrombosis
6. Pregnant woman
7. HIV positive

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2007-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Infection resolution rates within 5 days of treatment | 5 days (120 hours)
  PMN < 250/mm3 from ascitic fluid

SECONDARY OUTCOMES:
Mortality & recurrence rates within 1 month | 1 month
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Soon Ho Um, Professor, Principal Investigator — Korea University
Locations (2):
- South Korea (2):
  - Korea University Ansan Hospital, Ansan
  - Korea University Anam Hospital, Seoul

REFERENCES:
- [Derived] Yim HJ, Kim TH, Suh SJ, Yim SY, Jung YK, Seo YS, Kang SH, Kim MY, Baik SK, Kim HS, Kim YS, Park SY, Kim BI, Park JY, Heo J, Sohn JH, Heo NY, Han KH, Um SH. Response-Guided Therapy With Cefotaxime, Ceftriaxone, or Ciprofloxacin for Spontaneous Bacterial Peritonitis: A Randomized Trial: A Validation Study of 2021 AASLD Practice Guidance for SBP. Am J Gastroenterol. 2023 Apr 1;118(4):654-663. doi: 10.14309/ajg.0000000000002126. Epub 2023 Jan 3. PMID 36594820